CLINICAL TRIAL: NCT00033423
Title: Phase I, Multicenter, Open Label, Dose Escalation Of 90Y-Zevalin Radioimmunotherapy Using A Modified Treatment Regimen For Relapsed Or Refractory CD20+ B-Cell (Follicular/Transformed) Non-Hodgkin's Lymphoma
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069282; UAB-0127; UAB-F010806018; NCI-G02-2053
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): First radiation dose regimen of yttrium Y 90 ibritumomab tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan
- Cohort II (Experimental): Second radiation dose regimen of yttrium Y 90 ibritumomab tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan
- Cohort III (Experimental): Third radiation dose regimen of yttrium Y 90 ibritumomab tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan
- Cohort IV (Experimental): Fourth radiation dose regimen of yttrium Y 90 ibritumomab tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan
- Cohort V (Experimental): MTD radiation dose regimen of yttrium Y 90 ibritumomab tiuxetan
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 ibritumomab tiuxetan when administered in combination with rituximab in patients with relapsed or refractory low-grade, follicular, or transformed CD20-positive B-cell non-Hodgkin's lymphoma (NHL).
* Determine the toxicity of different doses of yttrium Y 90 ibritumomab tiuxetan in patients treated with this regimen.
* Determine the frequency of reversal of bone marrow involvement with NHL in patients treated with this regimen.
* Determine the antitumor response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of yttrium Y 90 ibritumomab tiuxetan.

Patients receive rituximab IV once weekly on weeks 1-4. After 4 doses of rituximab, patients without bone marrow involvement and cellularity greater than 50% expected receive rituximab IV once weekly on weeks 6 and 7 and yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes with the final dose of rituximab (day 43).

Cohorts of 5-6 patients receive escalating dose of yttrium Y 90 ibritumomab tiuxetan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 4 of 5 or 3 of 6 patients experience dose-limiting toxicity.

Patients are followed at 6 and 12 weeks, every 2-3 months for 2 years, and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 6-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade, follicular, or transformed CD20-positive B-cell non-Hodgkin's lymphoma (NHL)
* Relapsed after prior chemotherapy OR chemotherapy-resistant disease
* Failed at least 1 prior chemotherapy regimen
* CD20-positive B-cell population in lymph nodes or bone marrow for International Working Formulation A (small lymphocytic lymphoma) and transformed NHL
* Bone marrow involvement with lymphoma less than 25% bilaterally
* No impaired bone marrow reserve defined as at least 1 of the following criteria:

  * Prior myeloablative therapies with bone marrow transplantation or peripheral blood stem cell rescue
  * Platelet count less than 100,000/mm3
  * Bone marrow cellularity no greater than 15%
  * Marked reduction in bone marrow precursors of one or more cell lines (e.g., granulocytic, megakaryocytic, or erythroid)
  * Failed prior stem cell collection
* No CNS lymphoma, chronic lymphocytic lymphoma, or HIV or AIDS-related lymphoma
* No diffuse small lymphocytic/marginal zone lymphoma with lymphocyte count greater than 5,000/mm^3
* No pleural effusion NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 19 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit greater than 30%
* Hemoglobin greater than 9.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No anti-murine antibody reactivity if prior exposure to murine antibodies or proteins
* No other primary malignancy
* No other serious nonmalignant disease or infection that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior radioimmunotherapy
* Prior rituximab allowed if more than 6 months to progression after an objective response
* At least 6 weeks since prior rituximab
* At least 3 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* Recovered from prior immunotherapy

Chemotherapy:

* See Disease Characteristics
* No prior fludarabine
* At least 3 weeks since prior anticancer chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No concurrent chemotherapy

Endocrine therapy:

* At least 3 weeks since prior anticancer endocrine therapy
* No concurrent high-dose systemic corticosteroids (e.g., 50 mg or more of prednisone as a single dose or 50 mg or less of prednisone for more than 6 doses)

Radiotherapy:

* No prior radiotherapy to more than 25% of active bone marrow (involved field or regional)
* At least 3 weeks since prior anticancer radiotherapy and recovered

Surgery:

* At least 4 weeks since prior surgery (except diagnostic surgery) and recovered

Other:

* No other concurrent anticancer therapy
* Concurrent oral anticoagulant therapy allowed if platelet count is at least 30,000/mm3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of yttrium Y 90 ibritumomab tiuxetan when administered in combination with rituximab in patients with relapsed or refractory low-grade, follicular, or transformed CD20-positive B-cell non-Hodgkin's lymphoma (NHL). | baseline through 4 years

SECONDARY OUTCOMES:
Determine the toxicity of different doses of yttrium Y 90 ibritumomab tiuxetan in patients treated with this regimen | baseline through 4 years
Determine the frequency of reversal of bone marrow involvement with NHL in patients treated with this regimen. | baseline through 4 years
Determine the antitumor response in patients treated with this regimen. | baseline through 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero-Torres, MD, CSU, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Forero-Torres A, Besh S, Knox S, et al.: Higher doses of Rituxan alter pharmacokinetics and biodistribution of Zevalin but may increase responses; a preliminary report of a phase I study of Zevalin using a modified treatment regimen for relapsed or refractory CD20+ B-Cell follicular/transformed non-Hodgkins lymphoma. [Abstract] Blood 102 (11 Pt 1): A-1483, 2003.